CLINICAL TRIAL: NCT00075153
Title: Quality of Life in Children With HIV Infection
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 1R01NR007975-01 (NIH); R01NR007975 (NIH)
Record Dates: First submitted 2004-01-02; First posted 2004-01-08 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: ADOLESCENCE; HIV INFECTION; PEDIATRIC AIDS; QUALITY OF LIFE; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize the quality of life (QOL) and longitudinal patterns of change in QOL outcomes in children and youth with HIV infection; to identify demographic, social, disease status, treatment, and health care utilization factors that predict longitudinal changes in outcomes; to develop a conceptual model that characterizes the effects of specific factors that predict longitudinal changes in QOL; and to characterize the influence of HIV symptoms on QOL outcomes in the domains of health perceptions, physical, psychological, and social role functioning.

DETAILED DESCRIPTION:
This is a Phase III study. This study will use national data available through a prospective, observational, longitudinal study of children and youth (n=1,993) from birth to 25 with HIV infection (Pediatric AIDS Clinical Trials Group Protocol 219/219C) to develop knowledge about the quality of life (QOL) and the factors that affect it in order to be able to implement effective nursing interventions and clinical programs to support and improve QOL in this vulnerable population of children.

ELIGIBILITY:
Inclusion criteria

* Children and youth with perinatally acquired HIV infection
* Enrolled in PACTG 219/219C
* Completed quality of life assessment

Exclusion criteria

--HIV exposed, not infected

Ages: 10 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and youth, from birth to 25 years, with perinatally acquired HIV infection enrolled in PACTG 219/219C
Sampling Method: Non-Probability Sample
Enrollment: 1993 (Actual)
Dates: Start 2001-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life assessment | 1999

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S. Storm, MSN, PhD, Principal Investigator — School of Nursing, Rutgers, The State University of New Jersey
Locations (1):
- University of Medicine and Dentistry of NJ, Newark, New Jersey, United States